CLINICAL TRIAL: NCT01798433
Title: A Prospective, Multi-center, Randomized Study to Evaluate the Optimal Strategy for Side Branch Treatment in Patients With Left Main Coronary Bifurcation Lesion
Brief Title: STRATEGY for Left Main Coronary Bifurcation Lesion II
Acronym: STRATEGY-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-12-039
Record Dates: First submitted 2013-02-11; First posted 2013-02-25 (Estimated); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Coronary Artery Disease
Keywords: Angioplasty; Transluminal; Percutaneous Coronary
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- One stent technique alone (Experimental): One stent technique alone for non-true LM bifurcation
  Interventions: Device: One stent technique alone
- One stent technique + Elective FKB (Experimental): One stent technique + Elective FKB for non-true LM bifurcation
  Interventions: Device: One stent technique + Elective FKB
- Provisional approach (Experimental): Provisional approach for true LM bifurcation
  Interventions: Procedure: Provisional approach
- Elective 2-stent (Experimental): Elective 2-stent for true LM bifurcation
  Interventions: Device: Elective 2-stent

INTERVENTIONS:
Device: One stent technique alone — One stent technique alone with drug-eluting stent
  Arms: One stent technique alone
Device: One stent technique + Elective FKB — One stent technique + Elective FKB with drug-eluting stents + balloon
  Arms: One stent technique + Elective FKB
Procedure: Provisional approach — Provisional approach with drung-eluting stents
  Arms: Provisional approach
Device: Elective 2-stent — Elective 2-stent with drug-eluting stents
  Arms: Elective 2-stent

SUMMARY:
In patients with unprotected left main (LM) true bifurcation lesion (cohort A), elective 2-stent strategy is superior to provisional strategy at preventing the occurrence of 12-month target lesion failure after percutaneous coronary intervention for bifurcation lesion.

In patients with unprotected LM non-true bifurcation lesion (cohort B), 1-stent technique with mandatory final kissing ballooning is superior to 1-stent technique without kissing ballooning at preventing the occurrence of 12-month target lesion failure after percutaneous coronary intervention for bifurcation lesion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20 years
2. Left main bifurcation lesion on coronary angiography
3. Significant myocardial ischemia Main vessel (left main coronary artery and left anterior descending artery) and/or side branch (left circumflex artery) diameter stenosis > 75%, or diameter stenosis 50-75% with angina and/or objective evidence of ischemia in the non-invasive stress test
4. Significant size of the main branch (left anterior descending artery) and side branch (left cirmflex artery) - The reference diameter of both branches ≥ 2.5 mm by visual estimation

Exclusion Criteria:

1. The patient has a known hypersensitivity or contraindication to any of the following medications: Heparin, Aspirin, Clopidogrel, Biolimus
2. Patients who have received DES implantation in the target lesion prior to enrollment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-03-18 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 12-month
  defined ad a composite of cardiac death, spontaneous MI or target lesion revascularization

SECONDARY OUTCOMES:
Cardiac death | 12-month
  All deaths were considered cardiac unless a definite non-cardiac cause could be established.
Angiographic in-segment restenosis rate | 9 months
  as measured by 9-month quantitative coronary analysis
Target vessel revascularization (TVR) | 12-month
  TVR was defined as repeat revascularization of the target vessel by PCI or bypass graft surgery.
Stent thrombosis | 12-month
  Stent thrombosis was assessed based on the definitions of the Academic Research Consortium as definite, probable, or possible stent thrombosis.
Myocardial infarction (MI) | 12-month
  MI was defined as elevated cardiac enzymes (troponin or MB fraction of creatine kinase, CK-MB) more than the upper limit of the normal value with ischemic symptoms or electrocardiography findings indicative of ischemia that was not related to the index procedure.
Target lesion revascularization (TLR) | 12-month
  TLR was defined as repeat PCI of the lesion within 5 mm of stent deployment or bypass graft surgery of the target vessel.
Periprocedural CK-MB elevation | the first 48 hours after PCI
  Periprocedural enzyme elevation was defined as a rise in CK-MB ≥3 times the upper normal limit after the index procedure.
Procedure success rate | the first 48 hours after PCI
Procedure time | immediate after PCI
Amount of contrast dye | immediate after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea